CLINICAL TRIAL: NCT02066103
Title: Broncho-Adventitial Delivery of Paclitaxel to Extend Airway Patency in Malignant Airway Obstruction Patients
Acronym: BROADWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercator MedSystems, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TSP0147; 5R42CA141907-03 (NIH)
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Malignant Airway Obstruction Secondary to Non-small Cell Lung Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel

SUMMARY:
Assess the safety and feasibility of local oncological drug delivery into the bronchial wall after recanalization of subjects with malignant airway obstruction. Safety and feasibility (technical success) will be assessed.

This localized delivery is intended as an adjunct therapy and all subjects will receive standard of care oncology therapy as determined by their treating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver, and renal function
* Scheduled to undergo bronchoscopy for malignant airway obstruction as standard medical care
* Pathologically confirmed, unresectable primary or recurrent non-small cell lung cancer
* Measurable disease with obstruction into the airway
* Pathologically confirmed, unresectable primary or recurrent non-small cell lung cancer
* Patients undergo recanalization procedure of tumor during bronchoscopy
* Investigator is able to insert and deploy the Blowfish Catheter into the airway after recanalization

Exclusion Criteria:

* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Pregnant or nursing female subjects, or female subjects of child bearing potential who refuse to take a pregnancy test prior to their enrollment in this study
* Uncontrolled infection
* Presence or recent history of any systemic disorder or conditions, such as:

  * uncontrolled hypertension
  * type 1 diabetes
  * severe pulmonary hypertension
  * acute kidney injury
  * stroke (within the last 6 month)
  * myocardial infarction (within the last 3 months)
* Individuals with neurological, mental or psychiatric disorders
* Concurrent participation in another study involving investigational drugs or investigational medical devices
* Other (non-cancer) disease not stabilized within 1 month before the Screening Visit
* Known hypersensitivity to paclitaxel, Cremophor EL, or iodinated contrast media
* Any serious, uncontrolled comorbidity or condition that an Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the patient Intraoperative Exclusion Criteria
* Use of pulmonary airway stents and/or ongoing or initiation of local external beam or brachytherapy radiation
* Any intraoperative complications that per the investigator's judgment increase the risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Treatment safety | 12 weeks
  Adverse Events (AEs), Serious Adverse Events (SAEs), and all Unanticipated Adverse Device Effects (UADEs)
Technical success | procedure day
  Device deployment and infusion success

SECONDARY OUTCOMES:
Airway patency improvements | 6 weeks
Quality of Life | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Raleigh, North Carolina

REFERENCES:
- [Derived] Yarmus L, Mallow C, Akulian J, Lin CT, Ettinger D, Hales R, Voong KR, Lee H, Feller-Kopman D, Semaan R, Seward K, Wahidi MM. Prospective Multicentered Safety and Feasibility Pilot for Endobronchial Intratumoral Chemotherapy. Chest. 2019 Sep;156(3):562-570. doi: 10.1016/j.chest.2019.02.006. Epub 2019 Feb 15. PMID 30776363